CLINICAL TRIAL: NCT05730920
Title: A Single-center, Randomized, Single-blind Pilot Study to Evaluate Intravenous Methadone Versus EXPAREL Erector Spinae Plane Blockade in Pediatric Subjects Undergoing Adolescent and Juvenile Idiopathic Scoliosis Correction
Brief Title: IV Methadone Vs EXPAREL Erector Spinae Plane Blockade in Pediatric Subjects Undergoing Idiopathic Scoliosis Correction
Acronym: AIMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Casey Stondell, MD (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor-Investigator, Dr. Casey Stondell, MD, Pediatric Anesthesiologist, Shriners Hospitals for Children
Organization: Shriners Hospitals for Children (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCA2205
Record Dates: First submitted 2023-01-25; First posted 2023-02-16 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Adolescent Idiopathic Scoliosis; Juvenile Idiopathic Scoliosis
Keywords: scoliosis; methadone; exparel; regional anesthesia; erector spinae plane block; pediatric
MeSH Terms: conditions — Scoliosis | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravenous (IV) Methadone (Active Comparator): Subjects will receive IV methadone 0.2 mg/kg (maximum dose 20mg) via an infusion pump over 15 minutes while undergoing continuous monitoring. Additional IV methadone may be given during the case per the anesthesiologist's discretion, but the total dose may not exceed 20mg.
  Interventions: Drug: Methadone
- Liposomal Bupivacaine (LB, Exparel) (Experimental): Subjects will receive four-point ESPB with an admixture of LB and 0.25% bupivacaine hydrochloride. The total LB dose will be 4mg/kg, max dose of 266mg, while the total dose of bupivacaine hydrochloride will be 2mg/kg.
  Interventions: Drug: Liposomal bupivacaine (LB, Exparel)

INTERVENTIONS:
Drug: Methadone — IV Methadone
  Arms: Intravenous (IV) Methadone
Drug: Liposomal bupivacaine (LB, Exparel) — LB and bupivacaine hydrochloride via erector spinae plane blocks
  Arms: Liposomal Bupivacaine (LB, Exparel)

SUMMARY:
The goal of this pilot study is to assess the feasibility of conducting a randomized controlled trial at a single institution comparing erector spinae plane blockade (ESPB) with liposomal bupivacaine (LB, Exparel) to intravenous (IV) methadone for managing pain in pediatric subjects undergoing adolescent and juvenile idiopathic scoliosis correction. Specifically, the goal is to enroll 15 subjects in each group and to complete data collection for all subjects. If this pilot study is successful, we plan to then design a larger scale study powered to compare specific outcomes between the two groups.

DETAILED DESCRIPTION:
Enrolled subjects will be randomized to one of two groups: one group will receive intra-operative IV methadone as the primary means of controlling post-operative pain while the other group will instead receive intra-operative erector spinae plane blocks (ESPB) with liposomal bupivacaine (LB, Exparel) and bupivacaine hydrochloride as the primary means of controlling postoperative pain. All other aspects of peri-operative management will be standardized. Subjects and the post-operative care team will be blinded to which intervention was performed in order to reduce bias. Upon discharge, subjects will receive a wearable activity monitor and a daily journal in order to record post-discharge data. Subjects will receive weekly phone calls for data collection and then will have a final in-person clinic visit, at which point participation in the study will conclude.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose parent(s) or guardian(s) has/have signed and dated the informed consent form (ICF) for the subject to participate in the study
* Patients with a diagnosis of juvenile idiopathic scoliosis (JIS) or adolescent idiopathic scoliosis (AIS) who will have posterior spinal fusion surgery
* Male or female patients 11 to less than 18 years of age on the day of surgery.
* American Society of Anesthesiologists (ASA) Class 1-2.
* Able to adhere to the study visit schedule and complete all study assessments.

Exclusion Criteria:

* Body mass index ≥35 at the time of screening
* Contraindication to regional anesthesia (e.g., abnormal coagulation, infection at site)
* Current opioid use at the time of screening
* Current diagnosis of chronic pain
* Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications
* Administration of liposomal bupivacaine (LB, Exparel)
* Subject/parent/guardian primary language other than English or Spanish
* Inability of patient to verbally express symptoms such as pain and side effects (as in moderate to severe developmental delay)
* A prolonged QTc on preoperative EKG (QTc longer than 450 milliseconds)
* History of Torsades de Pointes
* Renal or hepatic impairment
* Diagnosed active seizure disorder
* Any other condition that causes patient to be ineligible for surgery, i.e. pregnancy.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-09-21 (Actual)

PRIMARY OUTCOMES:
Successful Enrollment and Data Collection of 30 Subjects | 2 years
  Assess the feasibility of completing a prospective randomized trial pilot study comparing Erector Spinae Plane Blockade (ESPB) with liposomal bupivacaine (LB) to intravenous methadone at a single institution in two years

SECONDARY OUTCOMES:
Opioid Consumption | 2 years
  Assess whether there is a difference in post-operative opioid consumption between the two study groups. This will evaluated by converting all long-acting opioids to daily morphine equivalents per unit of weight.
Pain Scores | 2 years
  Assess whether there is a difference in post-operative pain scores between the two study groups. Visual analog scale (VAS) scores with a minimum of 0 and a maximum of 10 will be used where 0 is no pain and 10 is the worst pain imaginable
Length of Stay | 2 years
  Assess whether there is a difference in hospital length of stay between the two study groups

CONTACTS AND LOCATIONS:
Overall Officials: Casey Stondell, MD, Principal Investigator — Shriners Children's
Locations (1):
- Shriners Hospitals for Children, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No